CLINICAL TRIAL: NCT02404064
Title: Laparoscopic Appendectomy for Uncomplicated Appendicitis: Does Antimicrobial Prophylaxis Really Matter? Randomized Control Trial
Brief Title: Laparoscopic Appendectomy for Uncomplicated Appendicitis: Does Antimicrobial Prophylaxis Really Matter?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Dan Hershko, Profesor, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 134-14
Record Dates: First submitted 2015-03-15; First posted 2015-03-31 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Cefazolin; Cefotaxime; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antibiotics perioperative (Other): dose of perioperative antibiotics (cefamezin 1g IV; metronidazole 500 mg IV) This is the standard of care of the department
  Interventions: Drug: cefamezin 1g IV; Drug: metronidazole 500 mg IV
- placebo - No Antibiotics perioperative (Placebo Comparator): The intervention is No Antibiotics perioperative
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: cefamezin 1g IV — perioperative antibiotics (Cefamizin 1g IV; )
  Other Names: Cefotaxime
  Arms: Antibiotics perioperative
Drug: metronidazole 500 mg IV — perioperative antibiotics (metronidazole 500 mg IV )
  Other Names: falgyl
  Arms: Antibiotics perioperative
Drug: Placebo — No perioperative antibiotics
  Arms: placebo - No Antibiotics perioperative

SUMMARY:
To compare surgical site infection (SSI) rate in patients undergoing laparoscopic appendectomy for acute uncomplicated appendicitis and treated with single dose regime of antibiotics versus group of patients undergoing laparoscopic appendectomy without antibiotics treatment. Patient will be given either single dose of perioperative antibiotics or no antibiotics before surgery.

DETAILED DESCRIPTION:
Laparoscopic appendectomies are performed by one of the 6 institutional attending surgeons. US and/or abdominal CT scans are obtained as clinically necessary to make the diagnosis of appendicitis. All of the appendectomies are initiated laparoscopically. Postoperative orders are controlled via a standard electronic order set for all operations.

Patients found to have acute uncomplicated appendicitis at appendectomy will be randomized to either single dose of perioperative antibiotics /On the second post-operative day the patient who has no fever and tolerating a regular diet, will be discharged home without oral antibiotics. On the post-operative, day seven after surgery all patients will be examined in the outpatient clinic on the presence of surgical site infection. then will be followed for a 30 days after surgery .

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of acute appendicitis based on clinical examination, US and/or computed tomographic (CT) scan, and acute uncomplicated appendicitis at laparoscopic appendectomy.

Exclusion Criteria:

* Patients with a documented allergy to any of the medications in the trial.
* Those with an abscess identified by computed tomographic (CT) scan before surgery are not included in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
The main target-point of the study is surgical site infection (SSI), defined according to the Centers for Disease Control (CDC). | 30 Days
  Criteria for a superficial incisional SSI are an infection occurring at the incision site within 30 days after surgery that involved only the skin and subcutaneous tissue and at least one of the following:
  purulent drainage from the incision; an organism isolated from a culture of fluid from the superficial incision; incisional pain, tenderness, localized swelling, redness, or heat, and the wound was opened;

CONTACTS AND LOCATIONS:
Overall Officials: Dan Hershko, Professor, Principal Investigator — haemek medical center